CLINICAL TRIAL: NCT02823067
Title: Pruritus and Pemphigoid in Nursing Home Patients
Acronym: SSENIOR
Status: Completed | Type: Observational
Sponsor: M.F. Jonkman (Other)
Responsible Party: Sponsor-Investigator, M.F. Jonkman, MD PhD, University Medical Center Groningen
Organization: University Medical Center Groningen (Other)
Other Study IDs: NL56232.042.15; METc 2015/605 (Other: Medical Ethical Committee UMCG); NTR5843 (Registry Identifier: Nederlands Trial Register)
Record Dates: First submitted 2016-06-28; First posted 2016-07-06 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Pemphigoid; Pruritus
Keywords: Pemphigoid; Bullous pemphigoid; Pruritus; Senile pruritus; Neuropsychiatric symptoms
MeSH Terms: conditions — Pemphigoid, Bullous; Pruritus | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Nursing home patients: Nursing home patients aged 65 years or above. One extra blood sample of 10 ml will be taken during a routine venapunction for immunoserology testing.
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — One extra blood sample of 10 ml will be taken during a routine venapunction for immunoserology testing.

SUMMARY:
The primary objective of this observational study is to describe the prevalence of pruritus and pemphigoid in nursing home patients. Secondary outcomes are the relationships of demographic factors and medical risk factors with pemphigoid, including dementia and neuropsychiatric symptoms, medication use and Karnofsky score.

DETAILED DESCRIPTION:
Pruritus or itch is the most common skin symptom in elderly patients and is estimated to affect more than 30% of nursing home patients. Clinical and experimental evidence suggests pruritus in elderly patients may be linked to pemphigoid. Pemphigoid is the most common autoimmune skin blistering diseases and mainly affects the elderly. It is successfully treatable with systemic therapy. However, pemphigoid is often missed as a cause of pruritus in elderly patients (nonbullous cutaneous pemphigoid). Although nursing home patients and patients with dementia in particular have the highest risk for development of pemphigoid, no study has been performed in this population so far. Including serological screening for pemphigoid in the diagnostic evaluation of chronic pruritus in nursing home patients may lead to the diagnosis of pemphigoid. Furthermore, chronic itch may be an unrecognized cause of neuropsychiatric symptoms in nursing home patients with dementia.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient of a nursing home
* Age 65 years or above
* Subject or their official representatives have signed informed consent

Exclusion Criteria:

* Age below 65 years
* Subjects who do not have signed informed consent
* Receiving treatment with any systemic immunosuppressive agents
* Terminally ill patients with a life expectancy of less than 4 weeks

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population will consist of 126 nursing home patients aged 65 years or above, living in a nursing home of the University Network Care of the Elderly - UMCG.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Presence of pruritus | Day 1
  Presence and intensity of pruritus will be determined (hetero-)anamnestically with the Bullous Pemphigoid Disease Area Index (BPDAI) VAS score and derivative score for all subjects.
Detection of circulating pemphigoid specific IgG autoantibodies by indirect immunofluorescence on 1M salt-split human skin substrate | Day 1
  IgG autoantibodies with epidermal side staining of artificial split; positive/negative, staining intensity IgG 1+,2+,3+
Detection of circulating pemphigoid specific IgG autoantibodies by indirect immunofluorescence microscopy on monkey esophagus substrate | Day 1
  Anti-basement membrane zone IgG autoantibodies; positive/negative, staining intensity IgG 1+,2+,3+
Concentration of anti-BP180 NC16A IgG autoantibodies by ELISA | Day 1
  Anti-BP180 NC16A IgG index; U/mL, cut-off value 9 U/mL
Concentration of anti-BP230 IgG autoantibodies by ELISA | Day 1
  Anti-BP230 IgG index; U/mL, cut-off value 9 U/mL
Detection of circulating pemphigoid specific IgG autoantibodies by immunoblot of keratinocyte extract | Day 1
  Presence/absence of circulating IgG autoantibodies against BP180 (180kDa) or BP230 (230kDa)

SECONDARY OUTCOMES:
Age | Day 1
  For all subjects
Sex | Day 1
  For all subjects
Comorbidities | Day 1
  Presence/absence of comorbidities dementia, cerebrovascular accident, Parkinson's disease, other neurological disease or other diseases
Karnofsky Performance Scale | Day 1
  0% - 100%
Medication | Day 1
  Registration of medication use for all subjects
Neuropsychiatric symptoms | Day 1
  Neuropsychiatric Inventory - Nursing Home version in Dutch

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Jonkman, MD PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided